CLINICAL TRIAL: NCT04029792
Title: Pilot Study to Evaluate the Effect of the Consumption of the Combination of Plant Extracts (BSL_EP028) on Joint Mobility, Physical Performance and Vitality
Brief Title: Evaluation of a Combination of Plant Extracts (BSL_EP028) on Joint Mobility
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C028
Record Dates: First submitted 2019-07-22; First posted 2019-07-23 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-07

CONDITIONS: Joint Diseases
Keywords: Plant extract; Joint Mobility; Physical performance; Vitality
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of Plant Extracts (BSL_EP028) (Experimental): Volunteers will take twice at day for 8 weeks a capsule containing the combination of a plant extracts (BSL_EP028)
  Interventions: Combination Product: Combination of plant extracts (BSL_EP028)
- Placebo (Placebo Comparator): Volunteers will take twice at day for 8 weeks a capsule containing maltodextrin.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Combination of plant extracts (BSL_EP028) — Each participant will consume 2 capsules daily, in the morning and at night without any restriction in the diet nor in their habits of life.
  Arms: Combination of Plant Extracts (BSL_EP028)
Combination Product: Placebo — Each participant will consume 2 capsules daily, in the morning and at night without any restriction in the diet nor in their habits of life.
  Arms: Placebo

SUMMARY:
The aim of this trial is to study the effect of the combination of plant extracts (BSL_EP028) on joint mobility, physical performance and vitality in a group of healthy older adults who remit some joint discomfort. This is a preliminary study whose purpose is to gather information for future studies.

DETAILED DESCRIPTION:
The natural aging process involves several body changes that can affect to the mobility of subjects. Among them, those that affect the joints may have the greatest impact on mobility. With age, there is a progressive loss of the cartilage that covers the joints, as well as the synovial fluid, which in turn increases the stiffness of the ligaments and tendons that allow joint mobility, which implies a reduction in muscle tone and bone strength. This joint degeneration produces pain and discomfort, which leads to stiffness and restriction of movement. Therefore, and as a consequence of this loss of mobility, subjects decrease their physical performance, which can affect their mood and vitality. All of these may lead to a loss of quality of life and to an increase of the risk of future adverse health events, such as disability, institutionalization, hospitalization and the need for home medical care.

For all these reasons, and considering the increase in the ageing population worldwide, it seems relevant to develop new strategies to improve joint mobility, physical performance and vitality that are safe for the consumer, affordable and not associated with undesirable side effects. In this regard, natural plant extracts have been widely used as a traditional remedy to reduce joint pain, reduce fatigue and improve mood and physical performance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women that have joint discomfort (WOMAC score >20)

Exclusion Criteria:

* Consumption of pharmacological treatments on an ongoing basis that may affect joint mobility (chondroprotectors, corticoids and/or interarticular therapy or infiltrations).
* Having undergone surgery for osteoarthritis and/or having a diagnosis of degenerative osteoarthritis made by a rheumatologist/traumatologist
* Consuming nutritional supplements containing antioxidant substances
* Consumption of analgesics and/or anti-inflammatory drugs on a continuous and/or scheduled basis and will continue to do so during the study, even if they do not have pain.
* Being unable to perform the physical tests required in the study.
* Have an allergy to some component of the study product.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Total Score of the WOMAC (Western Ontario and McMaster. Universities Osteoarthritis index) test | 8 weeks
  It is a questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items)
  * Stiffness (2 items)
  * Physical Function (17 items) The higher the score, the higher the amount of pain, stiffness, and a high level of functional limitations

SECONDARY OUTCOMES:
SF-36 Vitality score | 8 weeks
  Vitality score measured by the The Short Form (36) Health Survey (0-100 scale, the higher score the higher vitality)
Physical activity measurement | 8 weeks
  Physical activity level will measure by the International Physical Activity Questionnaire (IPAQ). Results will be reported as MET minutes a week

OTHER OUTCOMES:
Evaluation of Knee Pain | 8 weeks
  Knee pain will evaluate by a Visual Analogue Scale (VAS), range 0 to 10, being 0 no pain and 10 the maximun pain
Evaluation of Hip Pain | 8 weeks
  Hip pain will evaluate by a Visual Analogue Scale (VAS), range 0 to 10, being 0 no pain and 10 the maximun pain
Timed Up and Go test | 8 weeks
  This test evaluates mobility and balance by measuring the time it takes a person to get up from a chair, walk three meters, turn around, walk to the chair, and sit.
30 sec Chair Stand test | 8 weeks
  This test evaluates the strength and endurance of the lower limbs by measuring the number of times a person can get up from a chair, with arms crossed at the chest, for 30 seconds.
Manual Dynamometry | 8 weeks
  Evaluates the grip strength of both hands
Evaluation of Muscular power and fatigue of the lower limbs | 8 weeks
  We evaluate the strength-velocity profile that the person has in the lower limbs through a linear encoder. It measures the speed of execution of a squat (extension of hips and knees) with three different loads.
Goniometric study | 8 weeks
  Evaluates the angles and ranges of movement of the hip joint (flexo-extension, abduction-adduction, internal-external rotation) and the femorotibial (flexo-extension).

CONTACTS AND LOCATIONS:
Overall Officials: Helios Pareja Galeano, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain